CLINICAL TRIAL: NCT03056300
Title: A Prospective, Multi-Center Evaluation of a Powered Vascular Stapler in Video-Assisted Thoracoscopic Lobectomies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ethicon, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ESC-14-006
Record Dates: First submitted 2017-01-26; First posted 2017-02-17 (Actual); Results first posted 2018-12-17 (Actual); Last update posted 2019-01-30 (Actual); Status verified 2019-01

CONDITIONS: Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Powered vascular stapler (Experimental): Video-Assisted Thoracoscopic Lobectomy with powered vascular stapler
  Interventions: Device: Video-Assisted Thoracoscopic Lobectomy with powered vascular stapler

INTERVENTIONS:
Device: Video-Assisted Thoracoscopic Lobectomy with powered vascular stapler — Powered Vascular Stapler used on vessels

SUMMARY:
The primary objective of this trial is to demonstrate the effectiveness of the powered vascular stapler for transection of the pulmonary artery (PA) and pulmonary vein (PV) during Video-Assisted Thoracoscopic Lobectomy.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects with a confirmed or suspected diagnosis of stage IA to stage IIB non-small cell lung cancer scheduled for lobectomy (Lung Cancer Staging per American Joint Committee on Cancer,7th Edition)7;
2. Subjects scheduled for VATS lobectomy in accordance with their institution's SOC;
3. Performance status 0-1 (Eastern Cooperative Oncology Group classification);
4. ASA score < 3;
5. No prior history of VATS or open lung surgery (on the lung in which the procedure will be performed);
6. Willing to give consent and comply with study-related evaluation and treatment schedule; and
7. 18-75 years of age (inclusive).

Exclusion Criteria:

1. Active (subject currently receiving systemic treatment) bacterial infection or fungal infection;
2. Systemic administration (intravenous or oral) of steroids, including herbal supplements that contain steroids (within 30 days prior to study procedure);
3. Uncontrolled diabetes mellitus;
4. End stage renal or liver disease;
5. History of severe cardiovascular disease;
6. FEV1% <50% or severe COPD;
7. Prior chemotherapy or radiation for lung cancer;
8. Scheduled concurrent surgical procedure other than diagnostic wedge resection followed by lobectomy (central venous access - e.g., port placement, mediastinoscopy with lymph node sampling, and VATS lymphadenectomy are allowed);
9. Robotic-assisted procedure;
10. Women who are pregnant or lactating at the time of screening;
11. Physical or psychological condition which would impair study participation;
12. The subject is judged unsuitable for study participation by the Investigator for any other reason;
13. Participation in any other investigational drug (within 30 days or 5 half-lives of an investigational drug) or device study; or
14. Unable or unwilling to attend follow-up visits and examinations.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2017-01-11 (Actual); Primary Completion 2017-05-26 (Actual); Study Completion 2017-05-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Keneng Chen, Principal Investigator — Peking University Cancer Hospital & Institute; Shugeng Gao, Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Services; Hu Jian, Principal Investigator — The first affiliated hospital Zhejiang University/Hangzhou; Li Jian, Principal Investigator — Beijing Friendship hospital/Hangzhou
Locations (1):
- Beijing Cancer Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: Yes

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment occurred from January 2017 to April 2017 across 4 sites.
Pre-assignment Details: This was a single-arm study where all enrolled patients would have their surgery performed using the powered vascular stapler.
Groups:
- Powered Vascular Stapler: All enrolled subjects who had surgery performed using the powered vascular stapler.
Period: Overall Study
Arm/Group | Powered Vascular Stapler
Started | 50
Completed | 47
Not Completed | 3
Not completed — Surgical reason per study protocol | 3

BASELINE CHARACTERISTICS:
Population: All enrolled subjects who had a procedure completed and provided data on the number of surgical interventions.
Arm/Group | Powered Vascular Stapler
Number analyzed (Participants) | 50
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: All enrolled subjects who had a procedure completed and provided data on the number of surgical interventions.
  years | 59.2 (8.2)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: All enrolled subjects who had a procedure completed and provided data on the number of surgical interventions.
  Participants
    Female | 28
    Male | 22
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: All enrolled subjects who had a procedure completed and provided data on the number of surgical interventions.
  Participants
    American Indian or Alaska Native | 0
    Asian | 50
    Native Hawaiian or Other Pacific Islander | 0
    Black or African American | 0
    White | 0
    More than one race | 0
    Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants] — Population: All enrolled subjects who had a procedure completed and provided data on the number of surgical interventions.
  Participants
    China | 50

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Intra-Operative Hemostatic Interventions
Description: Incidence of hemostatic interventions/procedures completed for intra-operative bleeding related to the transection of the PA and PV during VATS lobectomy with the use of powered vascular stapler (PVS) defined as bleeding detected and controlled intraoperatively (additional stapling, over-sewing, clip placement, compression, use of suture, sealant, and/or buttress, and/or use of energy); or bleeding that occurs intra-operatively requiring blood or blood product transfusion or an additional surgical procedure (e.g. conversion to open).
Time Frame: Intra-Operative
Population: All enrolled subjects who had a procedure completed and provided data on the number of surgical interventions
Measure: Number (95% Confidence Interval); unit: Percentage of vessel transections
Units Other Than Participants: Vessel Transections
Arm/Group | Powered Vascular Stapler
Number analyzed (Participants) | 50
Number analyzed (Vessel Transections) | 167
Percentage of vessel transections | 1.8 [0.4 to 5.2]

2. Primary Outcome: Post-operative Interventions or Procedures Related to Pulmonary Artery or Pulmonary Vein Bleeding
Description: Incidence of hemostatic interventions /procedures completed for post-operative bleeding related to the transection of the PA and PV during VATS lobectomy with the use of PVS:
  * Hemostasis intervention: bleeding that occurs post-operatively requiring blood or blood product transfusion or an additional surgical procedure (related to PA and PV transection).
  No hemostasis intervention is defined as no interventions needed for post-operative bleeding (related to PA and PV transection).
Time Frame: Post-op through 4 week follow-up
Population: All enrolled subjects in whom a procedure was started.
Measure: Number (95% Confidence Interval); unit: Percentage
Arm/Group | Powered Vascular Stapler
Number analyzed (Participants) | 50
Percentage | 0 [0.0 to 7.1]

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time informed consent was signed through the final study visit which occurred approximately four weeks after the surgery was performed.
Arm/Group | Powered Vascular Stapler
All-Cause Mortality (participants affected / at risk) | 0/50
Serious Adverse Events (participants affected / at risk) | 5/50
Other Adverse Events (participants affected / at risk) | 12/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Powered Vascular Stapler (N=50)
Acute myocardial infarction (Cardiac disorders) | 1 (1)
Chylothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Powered Vascular Stapler (N=50)
Pyrexia (General disorders) | 5 (5)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Chest discomfort (General disorders) | 1 (1)
Wound complication (Injury, poisoning and procedural complications) | 1 (1)
Blood albumin decreased (Investigations) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary air leakage (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Subcutaneous emphysema (Skin and subcutaneous tissue disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
This was a single arm study with a limited sample size.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2016-02-11): https://cdn.clinicaltrials.gov/large-docs/00/NCT03056300/Prot_000.pdf
  • Statistical Analysis Plan (2017-07-06): https://cdn.clinicaltrials.gov/large-docs/00/NCT03056300/SAP_001.pdf